CLINICAL TRIAL: NCT03954418
Title: Trans-placental Transport and Foetal Accumulation of Artificial Sweeteners
Brief Title: Transport of Artificial Sweeteners During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MM_PO_MP_2019
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2019-05

CONDITIONS: Pregnancy Related; Diabetes; IUGR
Keywords: Artificial sweeteners; Non-nutritive sweeteners; Caesarean section
MeSH Terms: conditions — Diabetes Mellitus | interventions — acetosulfame; Cyclamates; Aspartame; Sweetening Agents

STUDY DESIGN:
Intervention Model Description: We wish to conduct an interventional, open-label study in which 40 women undergoing planned caesarean section will be included. In the intervention-group divided between:
  10 women with IUGR-child, 10 women with diabetes, 10 healthy women. We will use a control group of 10 healthy women who will refrain from intake.
  The participants will drink an artificially sweetened soft drink 2 to 4 hours before planned c-section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants will drink an artificially sweetened drink 2-4 hours before elective caesarean section.
  Interventions: Dietary Supplement: Acesulfame K, cyclamate, saccharine, aspartame
- Control group (No Intervention): Participants in the control group will refrain from intake of artificial sweeteners.

INTERVENTIONS:
Dietary Supplement: Acesulfame K, cyclamate, saccharine, aspartame — Intervention group receives a combination of multiple artificial sweeteners
  Other Names: Artificial sweeteners
  Arms: Intervention group

SUMMARY:
With obesity on the rise worldwide more and more young women are also affected, leading to a higher prevalence of obese pregnant women and pregnant women with diabetes.

Children of these women are in risk of developing obesity during childhood which again leads to overweight during adult life resulting in life-style related diseases such as diabetes and cardio-vascular disease.

Overweight and diabetic women are currently advised to substitute sugar sweetened beverages with artificially sweetened beverages to lower caloric intake and avoid fluctuations in blood glucose to avoid complications during pregnancy for both mother and child.

Recent studies suggest that high intake of artificial sweeteners during pregnancy increases the risk of the child developing obesity. If this is indeed true, the current guidelines have the opposite of the wanted and children already in risk of overweight are exposed to extra risk.

To investigate if artificial sweeteners can affect the foetus, the investigators wish to examine whether artificial sweeteners can cross the placenta.

The study is a clinical trial in which 40 women will be enrolled. 30 participants will drink a diet soft drink 2 hours before a caesarean section and 10 controls will refrain from intake. After birth the investigators will obtain a blood sample from the mother and from the umbilical cord and a placental biopsy and measure the contents of artificial sweeteners. Furthermore, the investigators will obtain a sample of amniotic fluid to examine if the sweeteners are excreted into the amniotic fluid.

The results ultimately have the potential to change the current guidelines on diet for overweight and diabetic women during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean section
* Child with IUGR (10 subjects)
* Diabetes (10 subjects)
* Other reasons for caesarean section(10 healthy subjects in intervention + 10 healthy controls)

Exclusion Criteria:

* Acute caesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Mothers blood | Time of birth
  Concentration of artificial sweeteners in blood from the mother
Placenta | Time of birth
  Concentration of artificial sweeteners in placenta
Umbilical cord | Time of birth
  Concentration of artificial sweeteners in blood from umbilical cord
Amniotic fluid | Time of birth
  Concentration of artificial sweeteners in amniotic fluid

CONTACTS AND LOCATIONS:
Overall Officials: Per Ovesen, DMSc, Study Director — per.ovesen@clin.au.dk
Locations (1):
- Obstetrics and Gynecology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No